CLINICAL TRIAL: NCT05629312
Title: Effect of Interceptive Strategies on the Clinical Outcome of Maxillary Impacted Canines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S59030
Record Dates: First submitted 2022-11-16; First posted 2022-11-29 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-12

CONDITIONS: Tooth, Impacted
Keywords: Interceptive orthodontics; maxillary canines; maxillary expansion; Tooth extraction; deciduous tooth
MeSH Terms: conditions — Tooth, Impacted | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maxillary expansion (Experimental): All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm present also lack of space in the upper jaw and are treated with maxillary expansion
  Interventions: Procedure: Maxillary expansion
- Extraction of deciduous canines (Experimental): All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm present also lack of space in the upper jaw and are treated with extraction of deciduous canines
  Interventions: Procedure: Extraction of deciduous upper canines
- No intervention (No Intervention): All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm present also lack of space in the upper jaw and no intervention is performed
- Control (No Intervention): All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm do not present lack of space in the upper jaw and no intervention is performed

INTERVENTIONS:
Procedure: Maxillary expansion — The upper jaw is expanded with a removable expansion plate
  Arms: Maxillary expansion
Procedure: Extraction of deciduous upper canines — Both deciduous upper canines are extracted in this group
  Arms: Extraction of deciduous canines

SUMMARY:
This study aims to investigate the effect of 3 randomly applied interceptive measures (slow maxillary expansion, extraction of deciduous canines and no intervention) on maxillary canine impaction in patients with early mixed dentition and lack of space in the dental arch. Additionally, these groups are compared with a control group with adequate space. Patients with at least one impacted maxillary canine, presence of deciduous canines and absence of crossbite were included. The canine position is assessed by measuring five variables (sector of the canine cusp, canine to midline angle, canine to first premolar angle, canine cusp to midline distance, and canine cusp to maxillary plane distance) on 2 panoramic radiographs at 0 (T1) and 18 months (T2).

DETAILED DESCRIPTION:
The detailed information regarding methodology has been entered in following sections

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting at the intake consultation of the Department of Orthodontics of University Hospitals Leuven, Belgium from September 2016, with at least one maxillary permanent canine impaction are invited to participate. Canine impaction is diagnosed based on a panoramic radiograph, taken for standard evaluation of dental development and associated pathology. A maxillary canine is considered to be impacted when the canine to midline angle was ≥15° (Alqerban et al. 2014; Warford et al. 2003). Only impacted maxillary canines with incomplete root formation and with persisting deciduous canines are included.

Exclusion Criteria:

* presence of uni- or bilateral posterior dental crossbite,
* upper permanent canines showing root malformation, ankylosis or fully erupted,
* evidence of root resorption of adjacent teeth, previous orthodontic treatment,
* craniofacial syndromes,
* systemic disease that would impede orthodontic treatment/surgery and recent exposure to radiotherapy.
* large eruption follicles seen on the permanent canines

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cadenas, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willems G, Butaye C, Raes M, Zong C, Begnoni G, Cadenas de Llano-Perula M. Early prevention of maxillary canine impaction: a randomized clinical trial. Eur J Orthod. 2023 Jul 31;45(4):359-369. doi: 10.1093/ejo/cjad014. PMID 37266982

RESULTS

PARTICIPANT FLOW:
Groups:
- Maxillary Expansion: All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm present also lack of space in the upper jaw and are treated with maxillary expansion
  Maxillary expansion: The upper jaw is expanded with a removable expansion plate
- Extraction of Deciduous Canines: All included patients (in all arms) present (at least one) maxillary canine impaction.
  Patients in this arm present also lack of space in the upper jaw and are treated with extraction of deciduous canines
  Extraction of deciduous upper canines: Both deciduous upper canines are extracted in this group
Period: Overall Study
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Started | 22 | 18 | 16 | 28
Completed | 19 | 17 | 14 | 26
Not Completed | 3 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Information not different to that of Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control | Total
Number analyzed (Participants) | 19 | 17 | 14 | 26 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 17 | 14 | 26 | 76
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.16) | 9.1 (1.46) | 9.0 (1.23) | 9.7 (1.44) | 9.2 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 6 | 5 | 30
  Male | 8 | 9 | 8 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 19 | 17 | 14 | 26 | 76
Region of Enrollment [Count of Participants; unit: Participants] — Leuven, Belgium
  Participants
    Belgium | 19 | 17 | 14 | 26 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Definitive Upper Canines That Erupt Spontaneously up to 18 Months of Follow up
Description: Number of definitive upper canines that erupt spontaneously up to 18 months of follow up.
Time Frame: 18 months
Population: This outcome measure (number 1) analyzes the amount of maxillary canines that have erupted per studied group within 18 months of the start of trial. Each included participant has two upper canines, all of them were analyzed. The Outcome Measure Data Table describes how many erupted after 18 months from all analyzed canines.
Measure: Number; unit: number of canines
Units Other Than Participants: number of upper canine teeth
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (number of upper canine teeth) | 38 | 34 | 28 | 52
number of canines | 3 | 2 | 1 | 4

2. Primary Outcome: Number of Definitive Upper Canines That Erupt Spontaneously After 18 Months of Follow up
Description: Number of definitive upper canines that erupt spontaneously after 18 months of follow up..
Time Frame: After the first 18 months of follow up
Population: This outcome measure (number 2) analyzes the amount of maxillary canines that have erupted per studied group after 18 months of the start of trial. Each included participant has two upper canines, all of them were analyzed. The Outcome Measure Data Table describes how many erupted after 18 months from all analyzed canines.
Measure: Number; unit: number of canines
Units Other Than Participants: number of upper canine teeth
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (number of upper canine teeth) | 38 | 34 | 28 | 52
number of canines | 4 | 4 | 6 | 15

3. Secondary Outcome: Sector Where the Canine is Located
Description: The sector is the position where the canine overlaps with adjacent teeth in a panoramic radiograph. The distance between the dental midline and the premolars is divided in 5 equally large spaces (units or categories 0 to 4) defined as follows: 0 = normal position (the cusp of the definitive canine is at the primary canine), 1 = distal to the long axis of the lateral incisor, 2 = mesial to the long axis of the lateral incisor, 3 = distal to the long axis of the central incisor, or 4 = mesial to the long axis of the central incisor This outcome measurement refers to the change in the Sector category where the canine is located, measured on a panoramic RX
Time Frame: 18 months
Population: Mean change in sector unit (where the canine is located) during the study period (18 months) per group
Measure: Mean (95% Confidence Interval); unit: Change in sector unit
Units Other Than Participants: sector where the canine is located
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (sector where the canine is located) | 38 | 34 | 28 | 52
Change in sector unit | -0.22 [-0.43 to -0.01] | -0.15 [-0.33 to 0.03] | 0.11 [-0.22 to 0.43] | -0.10 [-0.23 to 0.02]

4. Secondary Outcome: Angulation of the Canine Towards the Dental Midline
Description: Change in the Angulation of the canine towards the dental midline, measured on a panoramic RX
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: Degrees
Units Other Than Participants: Upper canine teeth
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (Upper canine teeth) | 38 | 34 | 28 | 52
Degrees | -11.85 [-15.99 to -7.71] | -8.16 [-13.19 to -3.13] | -7.68 [-13.76 to -1.60] | -11.29 [-15.06 to -7.52]

5. Secondary Outcome: Angulation of the Canine Towards the First Premolar
Description: Change in the Angulation of the canine towards the first premolar
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: Degrees
Units Other Than Participants: Upper canine teeth
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (Upper canine teeth) | 38 | 34 | 28 | 52
Degrees | -2.27 [-5.92 to 1.38] | -3.13 [-6.78 to 0.53] | 0.08 [-4.70 to 4.86] | -2.57 [-6.88 to 1.73]

6. Secondary Outcome: Distance Between the Canine Cusp and the Midline
Description: Change in the Distance between the canine cusp and the midline
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: Upper canine teeth cusp
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (Upper canine teeth cusp) | 38 | 34 | 28 | 52
millimeters | 0.83 [-0.58 to 2.24] | 0.57 [-0.65 to 1.80] | -0.51 [-2.21 to 1.19] | 1.77 [0.14 to 3.41]

7. Secondary Outcome: Distance Between the Canine Cusp and the Occlusal Plane
Description: Chenge in the Distance between the canine cusp and the occlusal plane, measured on a
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: Upper canine teeth cusp
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Number analyzed (Upper canine teeth cusp) | 38 | 34 | 28 | 52
millimeters | -6.31 [-9.82 to -2.80] | -4.79 [-6.87 to -2.71] | -7.10 [-10.78 to -3.43] | -9.14 [-11.78 to -6.51]

8. Secondary Outcome: Need for Further Minor and/or Major Orthodontic Intervention
Description: Need for further minor and/or major orthodontic interventions
Time Frame: 18 months after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
Number analyzed (Participants) | 19 | 17 | 14 | 26
Participants
  Minor intervention | 8 | 2 | 0 | 5
  MAjor intervention | 4 | 9 | 7 | 2

ADVERSE EVENTS:
Time Frame: 3 years (18 months during trial period, 18 months after trial period)
Description: The interventions studies cannot cause mortality
Arm/Group | Maxillary Expansion | Extraction of Deciduous Canines | No Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17 | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/14 | 0/26
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/14 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05629312/Prot_SAP_000.pdf